CLINICAL TRIAL: NCT00101062
Title: Phase II Study of Letrozole (Femara) and Celecoxib (Celebrex) in Postmenopausal Women With Hormone Receptor-Positive Locally Advanced or Metastatic Breast Cancer
Brief Title: Letrozole and Celecoxib in Treating Postmenopausal Women With Locally Advanced or Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: study drug unavailable
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Antionette Tan, MD, UMDNJ/CINJ
Organization: Rutgers, The State University of New Jersey (Other)
Masking: None | Purpose: Treatment
Other Study IDs: 040402-4671; CDR0000407502; P30CA072720 (NIH); CINJ-NJ1103; CINJ-5076v3; CINJ-040402; UMDNJ-4761
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Breast Cancer
Keywords: stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Celecoxib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: celecoxib
Drug: letrozole

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Hormone therapy using letrozole may fight breast cancer by lowering the amount of estrogen the body makes. Celecoxib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving letrozole with celecoxib may kill more tumor cells.

PURPOSE: This phase II trial is studying how well letrozole and celecoxib work in treating postmenopausal women with locally advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in postmenopausal women with hormone receptor-positive locally advanced or metastatic adenocarcinoma of the breast treated with letrozole and celecoxib as first-line therapy.

Secondary

* Determine the time to disease progression and overall survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Compare cyclooxygenase activity in blood and tumor cells from these patients before and after treatment with this regimen.
* Determine the effect of this regimen on aromatase activity, tumor proliferation, and angiogenesis in tumor samples from these patients.

OUTLINE: This is a multicenter study.

Patients receive oral letrozole once daily and oral celecoxib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 45-72 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the breast

  * Locally advanced or metastatic disease
* Measurable disease

  * No bone disease only
* No history of brain metastases unless controlled with radiotherapy or surgical resection for ≥ 6 months before study entry
* Hormone receptor status:

  * Estrogen receptor- OR progesterone receptor-positive

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Postmenopausal, as defined by 1 of the following:

  * Prior bilateral oophorectomy
  * Prior bilateral ovarian irradiation
  * No spontaneous menstrual bleeding within the past 12 months
  * Age 55 and over AND prior hysterectomy without oophorectomy
  * Age 54 and under AND prior hysterectomy without oophorectomy (or status of ovaries is unknown) AND documented follicle-stimulating hormone level in postmenopausal range

Performance status

* ECOG 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Granulocyte count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN

Other

* No prior allergic reaction attributed to compounds of similar chemical or biologic composition to study drugs
* No prior allergic reaction to sulfonamides
* No active peptic ulcer disease
* No active infection
* No other medical condition that would preclude study participation
* Able to swallow oral medication

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for metastatic or recurrent disease

Endocrine therapy

* No prior endocrine therapy for metastatic disease

  * Prior adjuvant tamoxifen allowed
* No prior aromatase inhibitors
* No prior hormonal therapy for recurrent disease
* No other concurrent hormonal therapy

Radiotherapy

* See Disease Characteristics
* See Menopausal status
* No concurrent radiotherapy

Surgery

* See Disease Characteristics
* See Menopausal status

Other

* No concurrent fluconazole or lithium
* No concurrent aspirin, non-steroidal anti-inflammatory drugs, or other cyclooxygenase-2 inhibitors

  * Concurrent chronic cardioprotective low-dose aspirin allowed
* No other concurrent investigational agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-01; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette R. Tan, MD, Study Chair — Rutgers Cancer Institute of New Jersey
Locations (1):
- Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://clinicaltrials.gov/ct2/show/NCT00101062